CLINICAL TRIAL: NCT01590355
Title: A Phase II Randomized Trial for Early-stage Squamous Cell Carcinoma of the Oropharynx: Radiotherapy vs Trans-oral Robotic Surgery (ORATOR)
Acronym: ORATOR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, David Palma, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORATOR
Record Dates: First submitted 2012-05-01; First posted 2012-05-02 (Estimated); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Early-Stage Squamous Cell Carcinoma of the Oropharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy; Neck Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiotherapy plus or minus Chemotherapy (Active Comparator): Radiotherapy plus or minus chemotherapy with surgical treatment for salvage of persistent disease
  Interventions: Radiation: Radiotherapy
- Transoral Robotic Surgery + Neck Dissection (Experimental): Transoral robotic excision will be carried out using the da Vinci surgical robot. The spatula cautery will be used to remove the tumours with 1 cm margins. At the time of surgery circumferential margins will be taken and sent for frozen section analysis. The resection will proceed until negative margins are obtained if feasible.
  Interventions: Procedure: Transoral Robotic Surgery + Neck Dissection

INTERVENTIONS:
Radiation: Radiotherapy — Gross Tumour and Nodes: 70 Gy in 35 fractions over 7 weeks. High-risk nodal areas: 63 Gy in 35 fractions over 7 weeks. Low-risk nodal areas: 56 Gy in 35 fractions over 7 weeks
  Arms: Radiotherapy plus or minus Chemotherapy
Procedure: Transoral Robotic Surgery + Neck Dissection — Transoral robotic excision will be carried out using the da Vinci surgical robot.
  Arms: Transoral Robotic Surgery + Neck Dissection

SUMMARY:
The historical standard treatment for early-stage squamous cell carcinoma of the oropharynx is radiation therapy. Some patients require chemotherapy with the radiation, and some patients require surgery if the tumour or lymph nodes have not responded after radiation.

This study will compare radiation therapy with a new surgical treatment called transoral robotic surgery (TORS). TORS is a new surgical approach using a robot to assist the surgeon in removing the tumour, potentially with fewer side effects than older surgical techniques.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* willing to provide informed consent
* ECOG performance status 0-2
* Histologically confirmed squamous cell carcinoma primary rumour site in the oropharynx (includes tonsil, soft palate, base of tongue, walls of oropharynx)
* Tumour stage:T1 or T2, with likely negative resections at surgery
* Nodal stage: N0, N1, or N2 (less than or equal to 4 cm in maximum dimension in any plane, on either side of the neck), without extranodal extension on pre-randomization imaging.
* Patient assessed at head and neck multidisciplinary clinic (with assessment by radiation oncologist and surgeon) and presented at multidisciplinary tumour board prior to randomization.

Exclusion Criteria:

* Serious medical comorbidities or other contraindications to radiotherapy, chemotherapy or surgery
* Prior history of head and neck cancer within 5 years
* Prior head and neck radiation at any time
* Metastatic disease
* Inability to attend full course of radiotherapy or follow-up visits
* Neck disease with unknown primary site
* Prior invasive malignant disease unless disease-free for at least 5 years or more, with the exception of non-melanoma skin cancer
* unable or unwilling to complete QoL questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-06; Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | 1-year post treatment

SECONDARY OUTCOMES:
Overall Survival | At the end of 3 years and at the end of 5 years
Progression-free survival | At the end of 3 years and at the end of 5 years
Quality of life at other time points | Every 6 months for 5 years from 1st date of treament
Toxicity | 5 years from date of first treatment
Swallowing Function | 5 years from date of first treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Palma, MD, PhD, Principal Investigator — London Regional Cancer Program of the Lawson Health Research Institute; Anthony Nichols, MD, Principal Investigator — London Regional Cancer Program of the Lawson Health Research Institute
Locations (6):
- Royal Adelaide Hospital, Adelaide, Australia
- Canada (5):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Nichols AC, Theurer J, Prisman E, Read N, Berthelet E, Tran E, Fung K, de Almeida JR, Bayley A, Goldstein DP, Hier M, Sultanem K, Richardson K, Mlynarek A, Krishnan S, Le H, Yoo J, MacNeil SD, Winquist E, Hammond JA, Venkatesan V, Kuruvilla S, Warner A, Mitchell S, Chen J, Johnson-Obaseki S, Odell M, Corsten M, Parker C, Wehrli B, Kwan K, Palma DA. Radiotherapy Versus Transoral Robotic Surgery for Oropharyngeal Squamous Cell Carcinoma: Final Results of the ORATOR Randomized Trial. J Clin Oncol. 2024 Dec;42(34):4023-4028. doi: 10.1200/JCO.24.00119. Epub 2024 Sep 20. PMID 39303189
- [Derived] Nichols AC, Theurer J, Prisman E, Read N, Berthelet E, Tran E, Fung K, de Almeida JR, Bayley A, Goldstein DP, Hier M, Sultanem K, Richardson K, Mlynarek A, Krishnan S, Le H, Yoo J, MacNeil SD, Winquist E, Hammond JA, Venkatesan V, Kuruvilla S, Warner A, Mitchell S, Chen J, Corsten M, Johnson-Obaseki S, Odell M, Parker C, Wehrli B, Kwan K, Palma DA. Randomized Trial of Radiotherapy Versus Transoral Robotic Surgery for Oropharyngeal Squamous Cell Carcinoma: Long-Term Results of the ORATOR Trial. J Clin Oncol. 2022 Mar 10;40(8):866-875. doi: 10.1200/JCO.21.01961. Epub 2022 Jan 7. PMID 34995124
- [Derived] Nichols AC, Theurer J, Prisman E, Read N, Berthelet E, Tran E, Fung K, de Almeida JR, Bayley A, Goldstein DP, Hier M, Sultanem K, Richardson K, Mlynarek A, Krishnan S, Le H, Yoo J, MacNeil SD, Winquist E, Hammond JA, Venkatesan V, Kuruvilla S, Warner A, Mitchell S, Chen J, Corsten M, Johnson-Obaseki S, Eapen L, Odell M, Parker C, Wehrli B, Kwan K, Palma DA. Radiotherapy versus transoral robotic surgery and neck dissection for oropharyngeal squamous cell carcinoma (ORATOR): an open-label, phase 2, randomised trial. Lancet Oncol. 2019 Oct;20(10):1349-1359. doi: 10.1016/S1470-2045(19)30410-3. Epub 2019 Aug 12. PMID 31416685
- [Derived] Nichols AC, Yoo J, Hammond JA, Fung K, Winquist E, Read N, Venkatesan V, MacNeil SD, Ernst DS, Kuruvilla S, Chen J, Corsten M, Odell M, Eapen L, Theurer J, Doyle PC, Wehrli B, Kwan K, Palma DA. Early-stage squamous cell carcinoma of the oropharynx: radiotherapy vs. trans-oral robotic surgery (ORATOR)--study protocol for a randomized phase II trial. BMC Cancer. 2013 Mar 20;13:133. doi: 10.1186/1471-2407-13-133. PMID 23514246